CLINICAL TRIAL: NCT05786430
Title: Phase II Trial of Lazertinib+Pemetrexed/Carboplatin in Patients With EGFR Sensitizing Mutation Positive Recurrent or Metastatic Non-Small Cell Lung Cancer Failed to Prior Lazertinib (LUCAS)
Brief Title: Lazertinib+Pemetrexed/Carboplatin in Patients With EGFR Sensitizing Mutation Positive Recurrent or Metastatic Non-Small Cell Lung Cancer Failed to Prior Lazertinib
Acronym: LUCAS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Chang Gon Kim, Principal Investigator, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-1142
Record Dates: First submitted 2023-02-03; First posted 2023-03-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental)
  Interventions: Drug: Lazertinib/Pemetrexed/Carboplatin

INTERVENTIONS:
Drug: Lazertinib/Pemetrexed/Carboplatin — Combination of lazertinib 240 mg (80 mg, 3 tablets) and pemed-S + carboplatin. Once a day lazertinib 240 mg pemed-S: 500mg/m2 q3w carboplatin: AUC5 q3w (only administered up to 4 cycles)

SUMMARY:
This trial is Phase II Trial of Lazertinib+Pemetrexed/Carboplatin in Patients with EGFR Sensitizing Mutation Positive Recurrent or Metastatic Non-Small Cell Lung Cancer Failed to prior lazertinib.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent;

   1. A patient who voluntarily provided a written consent form before participating in a clinical trial;
   2. A patient who voluntarily provided written consent for genetic research for genetics and/or exploratory research
2. Age and gender

   1. Those over 20 years old
   2. Female patients should agree to use proper contraception and should not be breastfeeding, and for women of childbearing age, there should be evidence that pregnancy is negative before the start of administration or satisfies one of the following criteria for screening A woman who is over 50 years of age and has amenorrhea for at least 12 months after she stops all foreign hormone treatments Record of irreversible surgical infertility by hysterectomy, bilateral hysterectomy, or bilateral hysterectomy, tubal ligation is not allowed Women under the age of 50 remain in a state of amenorrhea for at least 12 months after stopping all foreign hormone therapy, and their luteinizing hormone (LH) and follicular-stimulating hormone (FSH) levels are within the range of menopause
   3. Male patients who have not undergone vasectomy must agree to blocking contraception, that is, the use of condoms, and are prohibited from providing sperm up to three months after the last clinical trial
3. Target disease a) Patients with locally progressive or metastatic non-small cell lung cancer identified histologically or cytologically b) Eastern Oncology Cooperative Group (ECOG) Performance Status 0~2 c) Patient with at least three months of life expectancy A patient with at least one measurable lesion according to RECIST v1.1 criteria (the area that has received previous local treatment cannot be a target lesion. However, if three months have passed since the previous local treatment and the progression of the lesion is confirmed, it can be regarded as a target lesion.) e) Patients with EGFR mutations identified before administration of Lazertinib (L858R, Exon 19 deletion mutations must be confirmed by record) f) Patients who fail Lazertinib treatment (including all of the following cases)

Patient using Lazertinib as the primary treatment - A patient using Lazertinib after failing one kind of first- and second-generation EGFR TKI (Gefitinib, erlotinib, afatinib)

Exclusion Criteria:

1. The following interventional treatment

   a) Patients who received cytotoxic anticancer drugs for the treatment of advanced non-small cell lung cancer within 14 days before the first administration of the drug for clinical trial (excluding EGFR TKI-based and targeted treatments) Patients who received local treatment within four weeks of the first administration of a clinical trial drug (e.g. major surgery, radiation therapy (excluding a limited range of high-purpose bone radiation therapy), hepatic arterioembolization, catheter artery chemoembolization, chemoembolization, high-frequency resection, percutaneous ethanol injection or refrigeration)

   * Note: Conventional bone-oriented radiation therapy must be done only for mitigation within a limited radiation area. It must be a short-term course according to the recommendations of the testing agency, and must be completed at least seven days before the first administration of a clinical trial drug.

   A patient who is currently receiving a drug or herbal supplement known as an inhibitor or induction of CYP3A4 or cannot be discontinued at least one week before the first administration of lazertinib Except for alopecia, toxic patients with previous treatments exceeding the unresolved CTCAE 2 grade at the time of initial administration of clinical trial drugs e) A patient with a history of using cytotoxic anticancer drugs with Palliative treatment
2. Medical history and current disease l) intracranial metastasis with symptoms or requiring treatment (it must be completed at least two weeks before the first injection date of a drug for clinical trial, if steroid treatment is required). If the training membrane metastasis is asymptomatic or mild, it can be registered at the judgment of the patient

   a) Intracranial bleeding with symptoms or needs treatment b) Past history of interstitial lung disease (ILD), pharmacogenetic ILD, radiation pneumonia requiring steroid treatment, or ILD with evidence of clinical activity c) Diseases determined to be significant by researchers, including a history of other malignant diseases except for non-small cell lung cancer within the last three years (exception: treated cervical epithelial cancer, differentiated thyroid cancer without lymph node metastasis, skin cancer other than lymph node metastasis), evidence of severe or uncontrolled systemic diseases, uncontrolled high blood pressure and bleeding; d) The following cardiovascular diseases

   - History of congestive heart failure (CHF) of Grade 3 or higher or heart arrhythmia requiring treatment according to the New York Heart Association Classification (NYHA) criteria

   History of unstable angina or myocardial infarction experienced within six months prior to the first administration of clinical trial drugs e) Test results of known human immunodeficiency virus (anti-HIV Ab) are positive Patients with hepatitis B (HBV) surface antigen (HBsAg) positive, hepatitis C antibody (anti-HCV) positive, and other clinically active infectious liver disease, e.g. patients with a history of HCV, can be registered if antiviral therapy is completed and subsequently recorded in a document that HCV RNA is below the minimum quantitative limit. In the case of HBsAg positive, in the case of a negative polymerase chain reaction to HBV DNA g) Intractable nausea and vomiting, gastrointestinal diseases, patients who cannot be taken orally, and absorption disorders that are deemed to interfere with the absorption of Lazertinib * However, if a colonectomy is performed and does not involve clinically meaningful absorption disorders according to the researcher's judgment, research registration is possible h) A known history of hypersensitivity in clinical trial drugs

   i) clinically significant chronic infection or major medical or mental illness j) In a case where it is determined based on the researcher's judgment that the patient should not participate in the clinical trial because the patient is unlikely to be able to comply with the clinical trial procedures, restrictions and requirements
3. Heart and clinical laboratory test criteria:

   1. Any of the following heart criteria:

      Based on QTc levels measured by electrocardiogram (ECG) equipment during screening, QT interval (QTc) correction average > 470 msec As long as the clinical significance of rhythm, conduction, or form on the ECG during the break. For example, full left angle blocking, 3 degree heart blocking, 2 degree heart blocking, PR interval > 250 msec All factors that increase the risk of QTc extension or arrhythmia, such as heart failure, hypokalemia, congenital QT extension syndrome, combination medication known to extend the QT interval, QT extension syndrome, or family history of unexplained sudden death under the age of 40.
   2. Inadequate bone marrow reserve or organ function identified by the following experimental figures:

ANC <1.0 x 109/L Platelet count <100 x 109/L Hemoglobin <80 g/L

* alanine amino transferase (ALT) > 5 x ULN
* Aspartic acid amino transferase (AST) > 5 x ULN Total bilirubin > 3 x ULN If the serum level exceeds 1.5 x ULN, the estimated cleaning rate measured using the institutional standard method (e.g., the value calculated by the Cockcroft & Gault equation) is less than 45ml/min

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival, PFS | End of trial (approximately 3 years)
  PFS is defined as the period from the date of administration of the first clinical trial drug to the progression of the disease or death for any reason.
  The progression-free survival period is analyzed for groups that can be evaluated for validity.

SECONDARY OUTCOMES:
Overall Survival, OS | End of trial (approximately 3 years)
  Overall Survival, OS The overall survival period (OS) is evaluated based on the date of administration of the drug for the first clinical trial and the state of survival at the time of analysis. The total survival period is defined as the period from the date of administration of the first clinical trial drug to the date of death regardless of the cause.
  The entire survival period is analyzed for the safety analysis group. The total duration of survival is presented in a graph of Kaplan-Meier. Summarize the number of events, median values (calculated in Kaplan Meier graphs), and the percentage of test subjects whose events have not occurred in the 6th, 12th, and 18th months. Death, survival tracking, tracking failures, and the number and percentage of test subjects who withdrew consent are properly summarized.
Objective Response Rate, ORR | End of trial (approximately 3 years)
  Objective Response Rate, ORR) ORR is defined as the percentage of test subjects whose confirmed response was (RECIST 1.1) at least one full response (Complete Response, CR) or partial response (Partial Response, PR) before evidence of disease progression appears.
  The objective response rate is summarized for groups that can be evaluated for validity. The objective response rate is presented with a 95% confidence interval on both sides (assuming a normal distribution).
Duration of Response, DoR | End of trial (approximately 3 years)
  Duration of response (Duration of Response, DoR) DoR is defined as the time of occurrence from the date on which a later confirmed reaction was first recorded to the date on which the disease progress was recorded or the date of death (the same as the date of occurrence of the PFS event). The start of the reaction is defined as the most recent visit date identified as the first visit response PR or CR. If the disease has not progressed after the test subject has reached the reaction, the duration of the reaction is calculated using the time of PFS intermediate amputation.
  The duration of the response is analyzed for the sub-group of subjects who are CR/PR whose best overall response is confirmed among the groups that can be evaluated for validity.
Disease Control Rate, DCR | End of trial (approximately 3 years)
  Disease control rate (Disease Control Rate, DCR) The disease control rate (DCR) is defined as the Best Overall Response (BOR), and the percentage of test subjects whose extracranial and intracranial responses are CR, PR, responding, or SD.
  The disease control rate is summarized for groups that can be evaluated for efficacy.
  The disease control rate is presented with a 95% confidence interval on both sides (assuming normal distribution).
Treatment failure pattern | End of trial (approximately 3 years)
  Treatment failure pattern (Treatment failure pattern) For the pattern of treatment failures, both intracranial disease progression (Intracranial progression) and non-cranial disease progression (Extracranial progression) are divided into progress and recorded and analyzed.
  Patterns of treatment failure and overall survival following locoregional failure or distant metastasis. It will be checked through RECIST every 8 weeks, confirmed as RECIST 1.1. Overall survival is analyzed in the safety analysis group. Overall survival is presented as a Kaplan-Meier graph.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Ryun Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No